CLINICAL TRIAL: NCT06011551
Title: HYDRAFIL-D: HYDRogel Augmentation For Intervertebral Lumbar Discs
Acronym: HYDRAFIL-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ReGelTec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGT-2000PS
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease (DDD)
Keywords: Intervertebral Disc; Nucleus Pulposus; Disc Augmentation
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Prospective, dual arm, randomized, controlled pivotal study
Who Masked: Participant
Masking Description: Single-blind (participants will be blinded to treatment assignment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Arm (Experimental): Group A: continued non-surgical conservative medical management plus a percutaneous hydrogel spinal implant delivered via the HYDRAFIL System (the HYDRAFIL implant) (the "Treatment Arm")
  Interventions: Device: The ReGelTec HYDRAFIL™ System; Other: Conservative Care Management
- Control Arm (Sham Comparator): Group B: continued non-surgical conservative medical management plus advancement of the HYDRAFIL System delivery needle to inside the skin in the direction of the target disc(s) but without contacting the muscle layer or deeper (the "Control Arm")
  Interventions: Other: Conservative Care Management

INTERVENTIONS:
Device: The ReGelTec HYDRAFIL™ System — The ReGelTec HYDRAFIL System is designed to deliver an injectable hydrogel implant (the HYDRAFIL implant) for the treatment of a degenerative lumbar disc.
  Arms: Treatment Arm
Other: Conservative Care Management — Conservative care management (including physical therapy and/or pain medication)
  Other Names: Non-surgical conservative medical management

SUMMARY:
A multi-center, prospective, dual arm, randomized, controlled pivotal study to evaluate the safety and effectiveness of the ReGelTec HYDRAFIL™ System.

DETAILED DESCRIPTION:
This pivotal study is designed to evaluate the safety and effectiveness of the ReGelTec HYDRAFIL System in subjects with axial chronic low back pain (CLBP) due to degenerative disc disease (DDD) who continue to have severe back pain and dysfunction after at least six (6) months of conservative care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 22 to 85 years, inclusive
* Subjects presenting with LBP greater than leg pain and symptoms of DDD of the lumbar region (L1- S1) of at least six (6) months duration
* Presence of one (1) or two (2) symptomatic disc(s) (i.e., only 1-level or 2-levels may be treated during the study) as determined by Discography
* Symptomatic disc(s) exhibiting Grade 4 to 8 degeneration on the modified Pfirrmann scale as determined by MRI
* Failure to have their symptoms resolve or reduce following at least six (6) months of conservative care (as defined in the body of the protocol)
* Psychosocially, mentally and physically able and willing to fully comply with this protocol including adhering to follow-up schedule and requirements and filling out forms
* English fluency
* Signed informed consent

Exclusion Criteria:

* History of or active systemic or local infection
* Any skin disease or inadequate tissue coverage at the site of the proposed injection
* Annular tear or defect that shows free contrast extravasation into the epidural space during or after Discography
* Presence of more than two (2) symptomatic discs presenting with pain confirmed during Discography
* Presence of extruded or sequestered disc herniation (i.e., disc extrusions or sequestrations) at the symptomatic level(s) or on adjacent levels
* Presence of wide annular fissures confluent with large disc protrusions at the symptomatic level(s)
* Epidural steroid injection, intradiscal injection, trigger point injection, facet or medial branch block within 60 days of enrollment
* Opioid medication usage >60 MME (morphine milligram equivalent)/day or increase in opioid use within 60 days of enrollment
* Evidence of Modic type 3 changes
* Subjects presenting with radicular pain greater than back pain or by history within the past six (6) months. Radicular pain is defined as nerve pain following a dermatomal distribution and that correlates with nerve compression on imaging. Note: somatic referred pain is allowed
* Evidence of neurogenic claudication due to spinal stenosis
* Subjects with any prior back surgery on the lumbar spine
* History of vertebral fractures in the lumbar spine
* Evidence of severe compression of cauda equina
* Evidence of spinal segmental instability (spondylolysis or spondylolisthesis: Grade >1), severe spinal canal stenosis, isthmus pathology, or scoliosis [Cobb angle >20 at the index level(s)]
* Subjects with arachnoiditis
* Subjects who are prisoners or wards of courts
* Subjects involved in active litigation including worker's compensation cases
* Subjects on chronic anticoagulation due to a bleeding disorder and unable to safely stop anticoagulants, or has taken anticoagulants within three (3) days prior to procedure
* Subjects with LBP of non-spinal or unknown etiology
* Subjects who have a history (in the last five (5) years) of substance abuse or chemical dependency (pharmaceuticals, illicit drugs, alcohol) or are current abusers (using definition criteria from the Diagnostic and Statistical Manual of Mental Disorders (DSM-V))
* Subjects who have major psychiatric disorders, such as major depression, bipolar disorder and schizophrenia, as defined by the DSM-V
* If female, subjects who are pregnant or are trying to become pregnant during the course of the trial (due to risks of additional radiation exposures)
* Failure to understand informed consent or inability or unwillingness to adhere to the study follow-up visit schedule or other protocol requirements
* Subjects having participated in any other clinical study within the last three (3) months, or are actively participating in any other clinical study, or have planned participation in any other clinical study during the course of this trial. Note: subjects must agree they will not participate in any other clinical study during the course of this trial
* Body Mass Index (BMI) >35 kg/m2
* Current smoker or nicotine and/or tobacco user
* Known allergy or hypersensitivity to any of the device materials
* Endocrine or metabolic disorder known to affect osteogenesis
* Insulin-dependent diabetes mellitus
* Inability to undergo X-ray, MRI, CT scans or other radiographic assessments, including Discography
* Any comorbid medical condition which, in the best judgement of the Investigator, would make the subject unsuitable for inclusion in the study or interferes with the proper assessment of safety or effectiveness (e.g., systemic disease)
* Subjects with any active malignancy or who have been previously diagnosed with a malignancy and have evidence of residual disease
* Any degenerative or neurological condition that would interfere with evaluation of outcomes or that may generate an unacceptable risk of failure or postoperative complications
* Chronic or acute renal and/ or hepatic impairment
* Evidence of severe osteoporosis. The SCORES/MORES will be utilized to screen if a DEXA scan is indicated. If SCORES/MORES value ≥ 6; then a DEXA scan is required. Severe osteoporosis is defined as DEXA T-score < 2.5 (spine or hip) or QCT T-score < 80mg/cubic cm

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint of Clinical Success | 12-month
  The primary endpoint is a single composite endpoint reflecting five study outcomes (function, SAEs, SSIs, intercurrent events, and radiographic findings). The individual subject's outcome will be considered a success if all of the criteria are met at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Beall, MD, Principal Investigator — Clinical Investigations LLC; Kasra Amirdelfan, MD, Principal Investigator — IPM Medical Group
Locations (12):
- United States (11):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Source Healthcare, Santa Monica, California
  - Boomerang Healthcare (IPM Medical Group), Walnut Creek, California
  - DBPS Research (The Denver Spine & Pain Institute), Greenwood Village, Colorado
  - Southwest Florida Pain Center, Port Charlotte, Florida
  - NRSA Group (Florida Spine & Pain Specialists), Riverview, Florida
  - Horizon Clinical Research (Southern Pain and Spine), Jasper, Georgia
  - Spine Institute of Louisiana (The Spine Network), Shreveport, Louisiana
  - Clinical Investigations, Edmond, Oklahoma
  - Precision Spine Care, Tyler, Texas
  - Virginia iSpine Physicians, Richmond, Virginia
- Beam Research (Beam Radiology), Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Company Website — https://regeltec.com/
- See also: HYDRAFIL-D Study Website — https://www.hydrafilstudy.com/